CLINICAL TRIAL: NCT04029350
Title: A Multi-center, One-arm, Phase II Trial of Anlotinib Combined With Osimertinib as the Second-line Treatment in Stage IIIb-IV NSCLC With Confirmed EGFRm and T790M.
Brief Title: Study of Anlotinib Combined With Osimertinib as Second-line Treatment in Stage IIIb-IV NSCLC With Confirmed EGFRm and T790M
Acronym: ALTN-03
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-03-II-01
Record Dates: First submitted 2019-07-21; First posted 2019-07-23 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Combined With Osimertinib (Experimental): Anlotinib 12 mg once a day from day 1 to 14 of a 21-day cycle. Osimertinib 80mg p.o, qd. It should be continued until disease progress or toxicity cannot be tolerated or patients withdraw consent.
  Interventions: Drug: Anlotinib Combined With Osimertinib

INTERVENTIONS:
Drug: Anlotinib Combined With Osimertinib — Anlotinib：12mg/capsule, take once when limosis in the morning. If patients suffer from AEs, they can get declined dosage (10mg or 8mg).
  Osimertinib：80 mg/tablet， per os (p.o.) daily. It should be continued until disease progression or intolerable toxicity or patients withdraw of consent.
  Other Names: A+T

SUMMARY:
Evaluate the efficacy and safety of Anlotinib combined with Icotinib as the second-line treatment in stage IIIb-IV NSCLC patients with sensitive EGFR and T790M mutations.

DETAILED DESCRIPTION:
Anlotinib Hydrochloride is a kind of innovative medicines approved by State Food and Drug Administration（CFDA:2011L00661） which was developed by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β and c-Kit.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, locally advanced and/or metastatic IIIB, IIIC or IV non-squamous NSCLC or recurrent non-squamous NSCLC (according to the 8th Edition of the AJCC Staging system).
2. Non-small cell lung cancer (NSCLC) with an activating EGFR mutation (exon 19 deletion, L858R point mutation, or any other mutation known to be associated with EGFR TKI sensitivity); presence of an activating EGFR mutation may be documented in tumor tissue or by plasma testing.
3. Locally confirmed T790M mutation determined from biopsy (preferred) or on circulating tumour DNA, documented in tissue, plasma or serum after disease progression on the most recent first- or second-generation EGFR TK treatment regimen.
4. 18-75years，ECOG PS：0-2，Life expectancy of more than 3 months，with measurable lesion ( RECIST1.1).
5. ≥1 target lesion that has not received radiotherapy in the past 3 months and can be accurately measured in at least 1 direction；Previously received radiation therapy, but the radiotherapy area must be <25% of the bone marrow area, and radiation therapy must have closed for at least≥4 weeks at the time of enrollment.
6. Main organs function is normal.
7. Signed and dated informed consent.
8. The woman patients of childbearing age must agree to take contraceptive methods during the research and within another 8 weeks after treatment. Pregnancy test (blood serum test or urine) should be done within 7 days before the research and the result should be negative.The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after treatment.

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma); Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer)
2. Non-small cell lung cancer (NSCLC) with an EGFR C797S mutation.
3. Prior treatment with a third-generation EGFR TKI (i.e. Rociletinib, Olmutinib、BPI-15086、BPI-7711、Osimertinib); Prior treatment with agents targeting the VEGF pathway, including bevacizumab and Anlotinib.
4. Treatment with an EGFR TKI (i.e. erlotinib, gefitinib or afatinib) within 8 days or approximately 5 x half-life, whichever is longer, of the first dose of study treatment；Patients may not be receiving any other investigational agents and may not have participated in a study of an investigational agent or using an investigational device within five half-lives of the compound or 3 months, whichever is greater
5. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2 platinum-therapy related neuropathy
6. Any factor that would preclude adequate absorption of Osimertinib and Anlotinib, including refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection
7. Patients with obvious brain metastases, cancerous meningitis, spinal cord compression, or with brain or pia mater disease. (patient with brain metastases who have completed treatment 28 days before and the symptoms are stable can be Enrolled, also should have no cerebral hemorrhage symptoms confirmed by brain MRI, CT or venography evaluation
8. Patients who planned to receive systemic anti-tumor therapy within 4 weeks prior to allocation or during the course of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or receiving the Mitomycin C 6 weeks prior to medication). Extra-field radiotherapy (EF-RT) was performed 4 weeks prior to allocation or restricted radiotherapy for assessing tumor lesions within 2 weeks prior to allocation
9. Patients with any severe and/or uncontrolled disease, including:

   1. Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] > 140 mmHg and/or diastolic blood pressure [DBP] > 90 mmHg despite antihypertensive medication)
   2. Mean resting corrected QT interval (Fridericia's correction formula [QTcF]) > 470 ms ms obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived corrected QT (QTc) value; Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block); Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval;
   3. Active or uncontrollable serious infection (≥CTC AE Level 2 infection)
   4. Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need to be treated with antiretroviral therapy
   5. Poor control of diabetes (fasting blood glucose [FBG]> 10 mmol/L)
   6. Urine routine test protein ≥++, and confirmed 24 hours urine protein> 1.0 g
10. Long-term unhealed wounds or fractures
11. Evidence of bleeding diathesis or coagulopathy (including clinically significant hemoptysis)
12. Patients with artery/venous thrombotic occurred within 12 months before allocation, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism
13. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
14. Patients with a history of psychotropic medicine abuse and cannot quit or have mental disorders
15. Respiratory syndrome (dyspnea≥CTC AE 2), severe pleural effusion, ascites, pericardial effusion
16. History of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation; active infection including hepatitis B (HBV DNA level ≥1000 copies /mL), hepatitis C and human immunodeficiency virus (HIV)
17. Has a history of malignant tumors. Except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone curative treatment and have no disease recurrence within 5 years after the start of treatment
18. History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD9291 (osimertinib) or Anlotinib
19. Patient was diagnosed with disease which will severely endanger the security of patients or influence the completion of this research; Judgment by the investigator that should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | each 42 days up to PD or death (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"

SECONDARY OUTCOMES:
OS（Overall Survival） | up to 24 months
  OS was defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
ORR（Objective Response Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
DCR（Disease Control Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Adverse Events | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Richeng Jiang, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (4):
- China (4):
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei Provincial People's Hospital, Shijiazhuang, Hebei
  - Shanxi Provincal Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
De-identified individul participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Background] Han B, Li K, Wang Q, Zhang L, Shi J, Wang Z, Cheng Y, He J, Shi Y, Zhao Y, Yu H, Zhao Y, Chen W, Luo Y, Wu L, Wang X, Pirker R, Nan K, Jin F, Dong J, Li B, Sun Y. Effect of Anlotinib as a Third-Line or Further Treatment on Overall Survival of Patients With Advanced Non-Small Cell Lung Cancer: The ALTER 0303 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2018 Nov 1;4(11):1569-1575. doi: 10.1001/jamaoncol.2018.3039. PMID 30098152
- [Result] Akamatsu H, Teraoka S, Morita S, Katakami N, Tachihara M, Daga H, Yamamoto N, Nakagawa K. Phase I/II Study of Osimertinib With Bevacizumab in EGFR-mutated, T790M-positive Patients With Progressed EGFR-TKIs: West Japan Oncology Group 8715L (WJOG8715L). Clin Lung Cancer. 2019 Jul;20(4):e492-e494. doi: 10.1016/j.cllc.2019.03.002. Epub 2019 Mar 19. PMID 31085043
- [Result] Saito H, Fukuhara T, Furuya N, Watanabe K, Sugawara S, Iwasawa S, Tsunezuka Y, Yamaguchi O, Okada M, Yoshimori K, Nakachi I, Gemma A, Azuma K, Kurimoto F, Tsubata Y, Fujita Y, Nagashima H, Asai G, Watanabe S, Miyazaki M, Hagiwara K, Nukiwa T, Morita S, Kobayashi K, Maemondo M. Erlotinib plus bevacizumab versus erlotinib alone in patients with EGFR-positive advanced non-squamous non-small-cell lung cancer (NEJ026): interim analysis of an open-label, randomised, multicentre, phase 3 trial. Lancet Oncol. 2019 May;20(5):625-635. doi: 10.1016/S1470-2045(19)30035-X. Epub 2019 Apr 8. PMID 30975627
- [Result] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Derived] Wang X, Li Z, Wang L, Liang Y, Huang C, Chen P, Huang D, Song X, Ding C, Wang C, Jiang R. Osimertinib plus anlotinib for advanced NSCLC with acquired EGFR T790M mutation: results from a multicenter phase II study with ctDNA analysis. BMC Med. 2025 Apr 15;23(1):223. doi: 10.1186/s12916-025-04044-8. PMID 40234867